CLINICAL TRIAL: NCT01020045
Title: Effect of HIV Infection and HAART on Bone Homeostasis
Brief Title: Effect of HIV Infection and Highly Active Antiretroviral Treatment (HAART) on Bone Homeostasis
Acronym: OPG-2
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Ighovwerha Ofotokun, Associate Professor of Medicine, Emory University
Other Study IDs: IRB00027210; R01AR059364-01 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infection; Osteopenia; Osteoporosis
Keywords: HIV; Osteopenia; Osteoporosis
MeSH Terms: conditions — HIV Infections; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-seropositive, HIV seronegative: No intervention - biologic samples were collected from both HIV positive and HIV negative subjects
- Treatment naive subjects: HIV-seropositive subjects naive to antiretroviral therapy. HIV-seronegative subjects otherwise healthy.

SUMMARY:
Advances in HAART have been a huge success story in the management of HIV infection. However, serious metabolic complications including osteoporosis and bone fractures are increasingly been seen with HAART, and the responsible mechanisms remain poorly elucidated.

The skeleton continually regenerates through homeostatic bone remodeling. Osteoclasts the cells responsible for bone resorption form under the influence of the key osteoclastogenic cytokine Receptor- Activator of NF-KB (RANKL). The osteoclastogenic and pro-resorptive activities of RANKL are moderated by its physiological decoy receptor osteoprotegerin (OPG). Increase in the ratio of RANKL to OPG accelerates the rate of osteoclastic bone resorption leading to osteoporosis.

The investigators' preliminary studies have now demonstrated that in an animal model of HIV/AIDS, the HIV-1 Transgenic rat, the development of osteoporosis is recapitulated as observed in human patients. Furthermore, the investigators found that B cell expression of OPG is significantly downregulated, concurrent with a significant upregulation in production of RANKL.

DETAILED DESCRIPTION:
The investigators hypothesize that "immunological disruption of B cell number and/or function, may play a key causal role in the bone loss associated with HIV/AIDS, by driving a "switch" from OPG production to overproduction of RANKL". The investigators propose to determine the role of perturbations in B and T cells on OPG and RANKL production and on bone turnover.

This is a cross-sectional analysis of changes in BMD (DXA), and B cell and T cell function in HIV seronegative/seropositive subjects matched by known risk factors for osteoporosis. Serum will be collected for quantitation of total OPG and RANKL, and for biochemical markers of bone turnover (CTx, and TRAP5b), specific and sensitive markers of osteoclast activity, and for osteocalcin and P1NP, specific and sensitive markers of bone formation by commercial ELISAs. Peripheral blood mononuclear cells (PBMC) will be isolated and total and percentage frequency and absolute number (/mL) of B cells (CD19+) and T cells (CD3) and their subsets (CD4 and CD8). B cells (CD19) and T cells (CD3 and CD4 and CD8) will be immunomagnetically purified and OPG and RANKL mRNA and protein production quantitated by RT-PCR and ELISA respectively. As a secondary endpoint, B cells will be fractionated into subsets based on differential expression of the markers CD10, CD21 and CD27 and OPG and RANKL production quantitated by in each subset by intracellular staining and FACS analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (sero-negative) volunteers and otherwise healthy treatment naïve HIV-1 sero-positive patient.
2. Age >30<50 years and segregated into age and gender ranges as described above in section 3.2 (15 subjects per stratification based on Power Test).
3. Ability and willingness of subject or legal guardian/representative to give written informed consent.
4. Antiretroviral naivety.
5. No CD4 T-cell counts requirement.
6. Absence of non-HIV related active immunological or bone disorders such as;

   * Bone marrow or organ transplantation
   * Inflammatory bowel disease (ulcerative colitis, crohn's disease)
   * Multiple Myeloma
   * Osteogenesis imperfect
   * Osteomalacia
   * Osteosarcoma
   * Paget's disease
   * Postmenopausal osteoporosis
   * Rheumatoid arthritis
   * Systemic lupus erythematosus
7. Laboratory values obtained within 90 days prior to study entry:

   * Hemoglobin >9.4 g/dl
   * Creatinine < 2 mg/dl
   * AST (SGOT) < 2 x ULN
   * ALT (SGPT) < 2 x ULN

Exclusion Criteria:

1. Physical or biochemical evidence or a medical history of malignancy.
2. Currently (within the past 8 weeks) taking any medication with known influence on the immune or skeletal system (e.g. immune modulation therapy, glucocorticoids, steroid hormones, bisphosphonates).
3. The patient is not fully ambulatory.
4. Pregnancy or breast feeding.

Exclusion criteria are primarily centered on immunological aspects with bone related aspects secondary. This is because in our model immunological function is proximal to bone function. Consequently, use of vitamin D or calcium supplementation will not be exclusion criteria, but will be added as covariates in our analysis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy (HIV sero-negative) volunteers and otherwise healthy antiretroviral treatment naïve HIV-1 sero-positive patients, age >18 years.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To correlate serum and B cell and T cell OPG and/or RANKL production in treatment-naïve HIV-infected patients, with indices of bone turnover and structure and with viral load. | During entry visit

CONTACTS AND LOCATIONS:
Overall Officials: Ighovwerha Ofotokun, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Program Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Result] Titanji K, Vunnava A, Sheth AN, Delille C, Lennox JL, Sanford SE, Foster A, Knezevic A, Easley KA, Weitzmann MN, Ofotokun I. Dysregulated B cell expression of RANKL and OPG correlates with loss of bone mineral density in HIV infection. PLoS Pathog. 2014 Nov 13;10(10):e1004497. doi: 10.1371/journal.ppat.1004497. eCollection 2014 Oct. PMID 25393853
- See also: Dysregulated B Cell Expression of RANKL and OPG Correlates with Loss of Bone Mineral Density in HIV Infection — http://journals.plos.org/plospathogens/article?id=10.1371/journal.ppat.1004497